## Consent Document

Official Title: Improving the Academic Performance of First-Grade Students with Reading and Math Difficulty

NCT Number: NCT03991234

Document Date: 03/14/2019

| Study Title: Improving the Acad | emic Performance of First | -Grade Students with Rea | ding and Math Difficulty; PI: Lym |
|---|---|---|---|
| Fuchs; Version Date: 3/14/19 | | | |
| Date: | | | |

Dear Parent/Guardian:

I am a faculty member at Vanderbilt University. This year, I am doing a research project at your child's school. The purpose of this project is to identify how schools can improve children's math and reading performance. This first-grade project has been approved by the Metropolitan-Nashville Public Schools' central office, and your child's teacher has agreed to participate in this project.

As part of this project, we will help your child's teacher administer a math test near the start of the school year in one whole-class session that lasts 30 minutes. Everyone in the class takes this test, and your child's teacher will use the information to help plan your child's instruction.

If you give permission for your child to participate in the Vanderbilt project, we will also use your child's scores on this test to help us decide if the project is a good fit for your child. We will make this decision based on whether it looks like your child **may** develop difficulty in math and reading. If your child scores low on the whole-class math test, we will give your child some other tests in an individual session that last 1 hour. On these tests, children name letters, name numbers, read words, answer math problems, explain what words mean, and solve puzzles. A graduate student, who is a research assistant on this project and experienced working with children your child's age, will administer the tests. By the end of October, we will let you know whether your child has been selected to participate.

If your child is selected to continue, the following activities will occur. First, your child's teacher will complete a form that tells us your child's age, gender, ethnicity, race, history of special education, years retained, English language services status, and your child's school system ID number (we will use this ID number to help us follow your child if he or she changes schools this year).

Your child's teacher will also complete forms that describe how well your child pays attention and how hard he/she works in class and what other tutoring your child receives at school. Also, we will obtain information from the district about whether your child receives subsidized lunch from the district. If your child is a non-native English speaker, your child's teacher will also give us his/her English-speaking scores on the school's test.

We will also give your child some tests in two more individual sessions, each 1 hour long. On these tests, answer questions about sounds in words, read words, answer math problems, solve puzzles, and remember words and numbers they hear. A research assistant on this project who is experienced working with children your child's age will administer the tests. Near the end of the year, a research assistant will test your child again, in one 45-minute small-group sessions and two 45-minute individual sessions. The tests ask children to solve puzzles, answer math problems, read words, and answer questions about stories they read.

For three out of every four children, we will provide individual tutoring. Some students will receive reading tutoring. Some will receive math tutoring. Some will receive reading and math tutoring.

**Institutional Review Board** 



Other students will continue in their classroom math and reading program without any change from us. To determine whether your child receives tutoring from us and whether that tutoring is in reading or math or reading and math, we will randomly assign children (like picking names out of a hat). We will let you know if your child receives tutoring and if yes, in what area. Tutoring will occur 3 times per week, 35 minutes each time, for 15 weeks and will be conducted by a research assistant who has experience working with children. Sessions will be scheduled with your child's teacher and take place during the regular school day. We will work with the teacher to schedule tutoring so your child does not miss important reading or math class time.

Throughout the project, we will watch for signs that your child does not wish to participate (like crying or uncooperative behavior). If we see this two separate times, we will no longer include your child in the study, and we will let you know. Also, to ensure that testing and tutoring are conducted correctly, we will audio record those sessions. Please note that your child's name will <u>not</u> appear anywhere on the recordings. After the recordings are checked for accuracy and saved onto a secure server at Vanderbilt, the tapes will be destroyed.

We will also provide teachers with the results of your child's math and reading tests to help the teacher teach more effectively. Also, if 90% of the consent forms are returned, whether or not parents agree for their children to participate, all children in the class will receive a free sticker or pencil. There are no plans to pay you for your child's participation.

This project may help children in two ways: by providing teachers with math and reading test information to help them plan more effective teaching programs and by providing some children with tutoring to help them become stronger in math or reading.

We see no risk associated with your child's participation. A possible inconvenience may be the time it takes your child to take the tests. Also, if you like, we will provide test results to you. If you would like test results, please complete that part of the form at the end of this letter. Otherwise, only your child's teacher and the research staff will have access to test scores.

No information or scores will be added to your child's school records, and reports will not identify any individual or school. Names will be removed from tests and replaced with identification numbers. Research records will be stored for 1 year in locked files at Vanderbilt. Efforts will be made to keep information in your child's research record private and confidential but absolute confidentiality cannot be guaranteed. Your child's information may be shared, for example, with the Vanderbilt University Institutional Review Board, the Federal Government Office for Human Research Protections, or the federal funding agency. This would happen only if your child or someone else is in danger or if we are required to do so by law. Vanderbilt may also provide this project's data to other research projects not listed in this letter. If data are shared, please be assured that no one will be able to figure out your child was part of this project. (There are no plans to pay you for such use or transfer of information.) Because this study is supported by the National Institutes of Health, the data we collect are protected by a Certificate of Confidentiality. This means that, in some cases, we cannot release study information even if it is requested through legal means. Disclosures you consent to in this document (sharing your child's academic scores with his/her teacher and sharing data for other research projects) are not protected (if data are shared for future research, no one will be able to figure out your child was part of this project). Note that disclosures you choose to make are not protected.

**Institutional Review Board** 



If you would like more information about your child's participation in this project, please call me at **615-343-4782**. Also, if you have general questions about giving consent or about your child's rights as a research participant, you may call the Vanderbilt Institutional Review Board at 615-322-2918.

If you decide not to have your child participate, please understand that nothing bad will happen. Also, if you decide to have your child participate but change your mind, nothing bad will happen. Also, if your child's teacher changes her/his mind about participating in this project, we will let you know that your child is no longer participating. Finally, if you agree to have your child participate, please understand that participation is voluntary. He/she may withdraw at any time or you may withdraw your child by calling me at the first number shown above.

Please complete the form below and return it (with the rest of this letter) to your child's classroom. We have provided two copies of this letter so you can keep one copy. Thank you very much.

| CONSENT FOR | |
|---|---|
| 1. Please check one of the following choices: | |
| YES, I give permission for my child, (child's name) | , |
| to participate in this project. I understand that my child's withdraw from the project at any time. | participation is voluntary and that he/she may |
| <b>IF YES</b> : What is your child's date of birth (month/ | What is your child's date of birth (month/date/year): |
| Is your child a girl or a boy? | |
| NO, I do not wish for my child, (child's name) | , to participate in this project. |
| Parent/Guardian Name | Date |
| Parent/Guardian Signature | School |
| 2. If you would like test results, please provide your telephone | or mailing address: |
| My telephone number: | |
| My U.S. mail address: | |

**Institutional Review Board** 



Sincerely,